CLINICAL TRIAL: NCT04859699
Title: Reopening Schools Safely and Educating Youth Research Study
Brief Title: Reopening Schools Safely and Educating Youth Research Study (ROSSEY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Linda Ko, Professor, School of Public Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00014531-A; 1OT2HD107544-01 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Absenteeism
Keywords: SARS-CoV-2; School re-opening; Rural communities; Risk communication
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This arm will include schools(n=7) and the enrolled families from those schools assigned as the control group, who will not receive the COVID-19 health education comic books and video intervention.
- COVID-19 Comic Books and Videos (Active Comparator): This arm will include schools (n=7) and enrolled families from those schools that are randomized to receive the health education with comic books and videos focused on the benefits of preventive measures for COVID-19.
  Interventions: Behavioral: COVID-19 Health Education Comic Books and Videos

INTERVENTIONS:
Behavioral: COVID-19 Health Education Comic Books and Videos — Comic books and videos will be shared with intervention students and their parents to provide education on COVID-19 topics such as masking, social distancing and COVID-19 testing
  Arms: COVID-19 Comic Books and Videos

SUMMARY:
The study has three aims and involves a clustered randomized controlled trial (RCT) where K-5 schools will be the unit of randomization. Aim 1 involves a qualitative assessment of rural Latino community's social, ethical, behavioral needs and resources for students to return to school and maintain onsite learning. Aim 2 includes a clustered RCT in schools. Aim 3 involves qualitative assessment of implementation outcomes of the Yakima School District (YSD) testing program and risk communication intervention with school stakeholders, parents, and children.

DETAILED DESCRIPTION:
OBJECTIVE:

Aim 1. Identify the rural Latino community's social, ethical, behavioral needs and resources for students to return to school and maintain onsite learning using qualitative assessments with school stakeholders, parents, and students.

Aim 2. Evaluate the effectiveness of risk communication on student attendance and participation in SARS-CoV-2 testing using a cluster randomized controlled trial (RCT) with two intervention arms: intervention (SARS-CoV-2 Risk Communication) and comparison (control group) arm.

Aim 3. Assess implementation outcomes of the Yakima School District testing program and risk communication intervention with school stakeholders, parents, and children guided by the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework.

OVERVIEW:

The study has three aims and involves a clustered randomized controlled trial (RCT) where K-5 elementary schools will be the unit of randomization. Aim 1 will involve conducting qualitative assessments with school stakeholders, parents and students to to assess social, ethical, cultural, and behavioral concerns related to COVID-19 in the community. This data will be used to guide the development of the risk communication strategies (e.g., comic books and videos). Aim 2 includes a clustered RCT conducted in Yakima School District elementary schools to evaluate the effect of risk communication on testing uptake. We will assess primary outcome on students; parent/guardian will provide informed consent through either an online, paper, or telephone process to enroll in the study. Following consent, parent/guardians of participants will receive instructions on study procedures and complete the enrollment questionnaire either via online, on paper, or over the telephone with a study staff member. If the students attend a school that is randomized into the intervention group, they will receive the risk communication as three comic books and their parents will receive two videos at regular intervals throughout the study in English and Spanish. The communication intervention will highlight benefits of and address barriers to preventative behaviors, SARS-CoV-2 testing, and COVID-19 vaccines. Participants in the comparison group will receive the risk communication comic books and videos at the end of the study as part of the delayed intervention. Secondary outcome measures will be assessed for one index child in all families who have children enrolled in the study.

To prepare for this large trial, the study will institute a pilot study conducting weekly novel coronavirus surveillance testing in one school during April - June 2021 to understand the implementation steps and the workflow of working with schools. The larger RCT trial will be implemented in 14 K-5 schools in Fall 2021 - Spring 2023 school year.

All students in the Yakima School District has access to the Yakima School District's COVID-19 static testing site. Screening and symptomatic testing will be available (but not mandated) to Yakima School District students through the static site. School attendance and SARS-CoV-2 test results on students enrolled in our research study will come from schools.

STUDY POPULATION:

The schools participating in the study come from an agricultural region of Washington state.

STUDY TIME PERIOD:

August 2021-March 2023.

STATISTICAL ANALYSES: The primary analysis will be based on the average number of onsite learning hours per week over the study period for each student. The data will be analyzed using a linear mixed effects model with district and randomization arm as fixed effects, and school and classroom within school as random effects. Analyses will test for any difference between the randomization arms using α = 0.05 and report the comparisons between arms.

STUDY OUTCOMES:

The primary outcome for children will be absenteeism (hours per week missing onsite learning).

The secondary outcome will be assessed in parent/child dyads. Parents will share their child's physical activity and emotional regulation; and will be assessed for perceived stress, COVID-related stress, and depressive symptomatology for parents.

ELIGIBILITY:
Inclusion Criteria:

* Participant attends or works in a participating school for at least 2 days/week.
* Participant must be willing to comply with all study procedures, including weekly online check-ins and phone interviews.
* Participant should have consistent and reliable Internet access, either by smart phone or computer.
* Participant must be comfortable speaking English or Spanish.
* Participant must be able to provide online informed consent and/or legal guardian assent.

Exclusion Criteria:

* Individuals unable to provide informed consent / assent, except in cases where the participant has an available legal authorized representative and/or parent
* Individuals who are incarcerated
* Individuals with conditions that may preclude or limit the participant's ability to comply with study procedures, according to the investigators
* Children who are wards of the state and who have clinically-diagnosed dementia, terminal (<5 years) illness, major psychiatric illness, severe hearing impairment, and inability to move, which will be assessed during the distribution of the study recruitment packets to families.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ko, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Pascoe KM, Bishop S, Ci X, Ramirez M, Perez G, Ibarra G, Garza L, Linde S, Duran MC, Chae HY, Quigley T, Hassell L, Garrison MM, Drain PK, Shah PD, Ko LK. Factors that shape COVID-19 pediatric vaccine decision-making in rural agricultural communities: A qualitative study. Vaccine. 2024 Dec 2;42(26):126389. doi: 10.1016/j.vaccine.2024.126389. Epub 2024 Oct 4. PMID 39368130
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249
- [Derived] Ramirez M, Shah PD, Chu HY, Garza L, Linde S, Garrison MM, Zhou C, Bishop S, Ibarra G, Ko LK. Reopening schools safely and educating youth (ROSSEY) study: Protocol for a community-based, cluster randomized controlled trial. Contemp Clin Trials. 2024 Apr;139:107480. doi: 10.1016/j.cct.2024.107480. Epub 2024 Feb 19. PMID 38382823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (Child and parent dyad) were recruited from Yakima School District elementary schools from January 17, 2022 and November 4, 2022.
Pre-assignment Details: Parent-child dyads were counted individually and the number of participants reflects each individual in the study. Some parents had more than one child (siblings) included in the study.
Units Other Than Participants: schools
Groups:
- Health Communication Strategy: This arm will include schools (n=7) and enrolled families from those schools that are randomized to receive the health education with comic books and videos focused on the benefits of preventive measures for COVID-19.
Period: Overall Study
Arm/Group | Control Group | Health Communication Strategy
Started | 524; 7 schools (Parent (n=217), Child (n=307; 217 Index, 90 sibling)) | 571; 7 schools (Parent (n=246), Child (n=325; 246 index, 79 sibling))
T2 Follow-up | 441; 7 schools (Parent (n=191), Child (n=250; 191 Index, 59 siblings)) | 525; 7 schools (Parent (n=217), Child (n=308; 217 index, 91 sibling))
T3 Follow-up | 454; 7 schools (Parent (n=209), Child (n=245; 209 index, 36 sibling)) | 482; 7 schools (Parent (n=186), Child (n=296; 186 index, 110 sibling))
Completed | 454; 7 schools (Parent (n=209), Child (n=245; 209 index, 36 sibling)) | 482; 7 schools (Parent (n=186), Child (n=296; 186 index, 110 sibling))
Not Completed | 70; 0 schools | 89; 0 schools

BASELINE CHARACTERISTICS:
Population: Consented kindergarten through 5th grade students and parents enrolled in participating school district; children includes index and siblings. Children in the intervention arm = 325 (246 index and 79 siblings); Children in the control group = 307 (217 index and 90 siblings).
Groups:
- Control Group: This arm will include schools and the enrolled families assigned as the control group, who will not receive the COVID-19 health education comic books and video intervention.
- Health Communication Strategy: This arm will include schools that are randomized to receive the health education with comic books and videos focused on the benefits of preventive measures for COVID-19.
  COVID-19 Health Education Comic Books and Videos: Comic books and videos will be shared with intervention students and their parents to provide education on COVID-19 topics such as masking, social distancing and COVID-19 testing
- Total: Total of all reporting groups
Arm/Group | Control Group | Health Communication Strategy | Total
Number analyzed (Participants) | 524 | 571 | 1095
Age, Customized [Count of Participants; unit: Participants] — Population: Row categories are divided by age and parent, child
  Participants
    <=18 Years: number analyzed (Participants) | 307 | 325 | 632
    <=18 Years: Child | 307 | 325 | 632
    <=18 Years: Parent | 0 | 0 | 0
    Between 18-65 Years: number analyzed (Participants) | 0 | 0 | 0
    Between 18-65 Years: Child | 0 | 0 | 0
    Between 18-65 Years: Parent | 0 | 0 | 0
    >=65 Years: number analyzed (Participants) | 0 | 0 | 0
    >=65 Years: Child | 0 | 0 | 0
    >=65 Years: Parent | 0 | 0 | 0
    Unknown or Not Reported: number analyzed (Participants) | 217 | 246 | 463
    Unknown or Not Reported: Child | 0 | 0 | 0
    Unknown or Not Reported: Parent | 217 | 246 | 463
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The total is divided between category and parent, child
  Participants
    Male: number analyzed (Participants) | 172 | 171 | 343
    Male: Child | 145 | 146 | 291
    Male: Parent | 27 | 25 | 52
    Female: number analyzed (Participants) | 322 | 369 | 691
    Female: Child | 161 | 179 | 340
    Female: Parent | 161 | 190 | 351
    Prefer not to Answer: number analyzed (Participants) | 3 | 2 | 5
    Prefer not to Answer: Child | 1 | 0 | 1
    Prefer not to Answer: Parent | 2 | 2 | 4
    Unknown or Not Reported: number analyzed (Participants) | 27 | 29 | 56
    Unknown or Not Reported: Child | 0 | 0 | 0
    Unknown or Not Reported: Parent | 27 | 29 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The total is divided between category and parent, child
  Participants
    Child: number analyzed (Participants) | 307 | 325 | 632
    Child: Hispanic or Latino | 242 | 267 | 509
    Child: Not Hispanic or Latino | 58 | 57 | 115
    Child: Unknown or Not Reported | 7 | 1 | 8
    Parent: number analyzed (Participants) | 217 | 246 | 463
    Parent: Hispanic or Latino | 143 | 167 | 310
    Parent: Not Hispanic or Latino | 40 | 45 | 85
    Parent: Unknown or Not Reported | 34 | 34 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The total is divided between category and parent, child
  Participants
    RACE (NIH/OMB) Child: number analyzed (Participants) | 307 | 325 | 632
    RACE (NIH/OMB) Child: American Indian or Alaska Native | 6 | 1 | 7
    RACE (NIH/OMB) Child: Asian American, Native Hawaiian or Other PI | 1 | 0 | 1
    RACE (NIH/OMB) Child: Black or African American | 1 | 1 | 2
    RACE (NIH/OMB) Child: White | 41 | 48 | 89
    RACE (NIH/OMB) Child: More than One Race | 4 | 7 | 11
    RACE (NIH/OMB) Child: Other | 5 | 0 | 5
    RACE (NIH/OMB) Child: Prefer Not to Answer | 7 | 0 | 7
    RACE (NIH/OMB) Child: Unknown or Not Reported | 242 | 268 | 510
    RACE (NIH/OMB) Parent: number analyzed (Participants) | 217 | 246 | 463
    RACE (NIH/OMB) Parent: American Indian or Alaska Native | 3 | 3 | 6
    RACE (NIH/OMB) Parent: Asian American, Native Hawaiian or Other PI | 0 | 1 | 1
    RACE (NIH/OMB) Parent: Black or African American | 1 | 2 | 3
    RACE (NIH/OMB) Parent: White | 35 | 36 | 71
    RACE (NIH/OMB) Parent: More than One Race | 1 | 3 | 4
    RACE (NIH/OMB) Parent: Other | 5 | 0 | 5
    RACE (NIH/OMB) Parent: Prefer Not to Answer | 9 | 0 | 9
    RACE (NIH/OMB) Parent: Unknown or Not Reported | 163 | 201 | 364
Region of Enrollment [Number; unit: participants] — Region of Enrollment Children
  participants
    United States | 307 | 325 | 632
Region of Enrollment [Number; unit: participants] — Region of Enrollment Parent
  participants
    United States | 217 | 246 | 463

OUTCOME MEASURES:

1. Primary Outcome: School Attendance
Description: How many school days missed due to symptoms of respiratory illness (only include index child).
Time Frame: Up to nine months
Population: Total number of school days missed by students (index child only) due to symptoms of respiratory illness at Post Survey 1 (Control = 191; Intervention = 217)
Measure: Mean (Standard Deviation); unit: Mean # days missed
Groups:
- COVID-19 Comic Books and Videos: This arm will include schools that are randomized to receive the health education with comic books and videos focused on the benefits of preventive measures for COVID-19.
  COVID-19 Health Education Comic Books and Videos: Comic books and videos will be shared with intervention students and their parents to provide education on COVID-19 topics such as masking, social distancing and COVID-19 testing
Arm/Group | Control Group | COVID-19 Comic Books and Videos
Number analyzed (Participants) | 191 | 217
Mean # days missed | 6.57 (7.72) | 7.34 (8.45)

2. Secondary Outcome: Emotional Regulation of Index Children at Baseline (T1)
Description: Index children will be assessed for physical activity, perceived stress, COVID-related stress, and depressive symptomatology from the PROMIS measures of Index Child Only (n=463) PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. PROMIS scores are typically reported on a T-score metric, with a mean of 50 and a standard deviation of 10. Higher T-scores indicate moderate to severe symptoms. T-scores above 60 are considered moderate, and those above 70 indicate severe symptoms.
Time Frame: Completed at baseline (T1)
Population: Overall ppts analyzed 463 index children, which is 217 at Control and 246 Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | COVID-19 Comic Books and Videos
Number analyzed (Participants) | 217 | 246
score on a scale
  Anxiety | 45.7 (9.65) | 45.4 (10.2)
  Stress | 49.2 (9.24) | 48.4 (9.07)
  Physical Activity | 48.8 (8.36) | 48.1 (8.02)
  Sleep Disturbance | 51.7 (10.0) | 51.0 (9.94)
  Depression | 43.9 (10.1) | 43.3 (9.76)

3. Secondary Outcome: Perceived Stress of Parents at Baseline (T1)
Description: Parents of enrolled children will be assessed for perceived stress, sleep disturbance, and emotional regulation using PROMIS measure.
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. PROMIS scores are typically reported on a T-score metric, with a mean of 50 and a standard deviation of 10. Higher T-scores indicate moderate to severe symptoms. T-scores above 60 are considered moderate, and those above 70 indicate severe symptoms.
  .
Time Frame: Completed at baseline (T1)
Population: Total number of Parents assessed for anxiety, sleep disturbance, depression, and stress
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | COVID-19 Comic Books and Videos
Number analyzed (Participants) | 217 | 246
score on a scale
  Anxiety | 52.6 (10.2) | 52.2 (10.6)
  Sleep distubance | 51.1 (9.73) | 50.5 (8.78)
  Depression | 48.4 (9.68) | 48.3 (10.1)
  Stress | 51.0 (8.51) | 51.0 (9.74)

4. Secondary Outcome: Emotional Regulation of Index Children at Post Survey 1 (T2)
Description: Post Survey assessment using PROMIS measures will evaluate physical activity, perceived stress, COVID-related stress, and depressive symptoms among 408 index children, out of an original cohort of 463, with 55 lost to follow-up. PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. PROMIS scores are typically reported on a T-score metric, with a mean of 50 and a standard deviation of 10. Higher T-scores indicate moderate to severe symptoms. T-scores above 60 are considered moderate, and those above 70 indicate severe symptoms.
Time Frame: Post survey 1 (T2)
Population: Overall ppts analyzed 408 index children, which is 191 at Control and 217 Intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | COVID-19 Comic Books and Videos
Number analyzed (Participants) | 191 | 217
score on a scale
  Anxiety | 45.9 (9.00) | 45.8 (10.0)
  Stress | 51.7 (8.97) | 51.7 (9.03)
  Physical Activity | 50.2 (7.46) | 50.1 (8.20)
  Sleep Disturbance | 52.6 (9.90) | 51.7 (10.5)
  Depression | 43.6 (9.50) | 42.4 (9.82)

5. Secondary Outcome: Perceived Stress of Parents at Post Survey 1 (T2)
Description: as for outcome 3
Time Frame: Completed at Post survey 1 (T2)
Population: Total number of Parents assessed for anxiety, sleep disturbance, depression, and stress
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | COVID-19 Comic Books and Videos
Number analyzed (Participants) | 191 | 217
score on a scale
  Anxiety | 53.1 (10.2) | 52.6 (10.5)
  Sleep distubance | 50.9 (9.25) | 49.2 (9.15)
  Depression | 48.9 (10.4) | 48.8 (10.2)
  Stress | 52.0 (10.2) | 51.0 (10.0)

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Description: Same as clinical trials
Groups:
- Control Group -Parent; Control Group - Child: This arm will include schools and the enrolled families assigned as the control group, who will not receive the COVID-19 health education comic books and video intervention.
- Health Communication Strategies Parent; Health Communication Strategies - Child: This arm will include schools that are randomized to receive the health education with comic books and videos focused on the benefits of preventive measures for COVID-19.
  COVID-19 Health Education Comic Books and Videos: Comic books and videos will be shared with intervention students and their parents to provide education on COVID-19 topics such as masking, social distancing and COVID-19 testing
Arm/Group | Control Group -Parent | Health Communication Strategies Parent | Control Group - Child | Health Communication Strategies - Child
All-Cause Mortality (participants affected / at risk) | 0/217 | 0/246 | 0/307 | 0/325
Serious Adverse Events (participants affected / at risk) | 0/217 | 0/246 | 0/307 | 0/325
Other Adverse Events (participants affected / at risk) | 0/217 | 0/246 | 0/307 | 0/325

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04859699/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04859699/SAP_001.pdf